CLINICAL TRIAL: NCT02616744
Title: A Single--blind, Randomized, Placebo--controlled Phase II Study to Evaluate the Impact of Oral Bisphosphonate Treatment on Bone Mineral Density in Osteopenic Women Receiving Adjuvant Aromatase Inhibitors - BONADIUV Trial
Brief Title: Study of Oral Bisphosphonate for Osteopenic Women Treated With Adjuvant Aromatase Inhibitors
Acronym: BONADIUV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BONADIUV
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitors; breast cancer; bone mineral density
MeSH Terms: conditions — Breast Neoplasms | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Ibandronic acid (Experimental): Ibandronic acid 150 mg per os per month for two years
  Interventions: Drug: Ibandronic acid
- Arm B: Placebo (Placebo Comparator): Placebo per os per month for two years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibandronic acid — 150 mg per month oral ibandronate
  Other Names: Ibandronate
  Arms: Arm A: Ibandronic acid
Drug: Placebo — 1 oral capsule of placebo per month
  Other Names: Placebo capsule
  Arms: Arm B: Placebo

SUMMARY:
A single--blind, randomized, placebo--controlled phase II study to evaluate the impact of oral bisphosphonate treatment on bone mineral density in osteopenic women receiving aromatase inhibitors as adjuvant treatment.

DETAILED DESCRIPTION:
Aromatase inhibitors (AIs) are the adjuvant treatment of choice in postmenopausal women with early, hormone receptor-positive breast cancer (BC), because they produce improved survival rates compared with tamoxifen. Progressive bone loss and subsequent fractures are associated with adjuvant AIs, administered either alone or sequentially after tamoxifen in postmenopausal women with early BC. Recent findings of National Surgical Adjuvant Breast and Bowel Project (NSABP) B-34 also suggest that bisphosphonates might have anticancer benefits for older postmenopausal women. "BONADIUV" trial is a single-blind, randomized, placebo-controlled study designed to evaluate the impact of bisphosphonate treatment on bone mineral density (BMD) in women taking AIs.

Patients undergo a baseline BMD and if they result osteopenic (lumbar spine and/or trochanter -1< T-score <2.5), they are randomized in a 1:1 ratio to receive either placebo or oral ibandronate. All patients receive oral supplementation of calcium and Vitamin D3, once daily for two years. Study duration is 2 year, with planned six-months evaluation.

A total of 72 patients per arm of treatment are needed to obtain a 85% statistical power in order to detect a 2% BMD mean difference between the two arms. Considering a 15% dropout, around 82 patients per arm are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hormone-receptor positive early breast cancer
* Menopausal status
* Age < 75 years
* Written informed consent

Exclusion Criteria:

* Premenopausal status at time of randomization
* Comorbidities with increased risk of osteoporosis (primary hyperparathyroidism, hyperthyroidism, rheumatoid arthritis)
* BMI < 18
* Chronic use of steroids
* Use of bisphosphonates at time of randomization
* Psychiatric disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lumbar spine and trochanter T-score mean difference as measure of BMD variation | 2 years
  Lumbar spine and trochanter T-score mean difference

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
  Number of Participants with Adverse Events
Overall Survival (OS) | 5 years
  Overall Survival (OS) rate
Disease-free Survival (DFS) | 5 years
  Disease-free Survival (DFS) rate

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Livi, Professor, Principal Investigator — AOU Careggi - University of Florence, Florence, Italy; Meattini Icro, M.D., Principal Investigator — AOU Careggi - University of Florence, Florence, Italy
Locations (1):
- Radiation Oncology Unit, Azienda Ospedaliero-Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Livi L, Scotti V, Desideri I, Saieva C, Cecchini S, Francolini G, Becherini C, Delli Paoli C, Visani L, Salvestrini V, De Feo ML, Nori J, Bernini M, Sanchez L, Orzalesi L, Bianchi S, Meattini I. Phase 2 placebo-controlled, single-blind trial to evaluate the impact of oral ibandronate on bone mineral density in osteopenic breast cancer patients receiving adjuvant aromatase inhibitors: 5-year results of the single-centre BONADIUV trial. Eur J Cancer. 2019 Feb;108:100-110. doi: 10.1016/j.ejca.2018.12.005. Epub 2019 Jan 14. PMID 30648627